CLINICAL TRIAL: NCT05472415
Title: Effects of Cognicise and Arch Support Insoles on Lower-extremity Function in Community-dwelling Older Adults With Mild Cognitive Impairment
Brief Title: Effects of Cognicise and Arch Support Insoles in Older Adults With Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, CY Song, Associate professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 110A-37
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): cognicise training with insole intervention
  Interventions: Other: cognicise; Device: arch support insoles
- control group (Active Comparator): cognicise training
  Interventions: Other: cognicise

INTERVENTIONS:
Other: cognicise — a combination of "cognition" and "exercise" training
Device: arch support insoles — The FootDisc insole is designed with curEVA for shock absorption and motion reduction, poron for secondary heel and metatarsal protection, and dynamic arch support for returning energy for propulsion
  Arms: experimental group

SUMMARY:
The purpose of this study aims to explore the surplus effect of arch support insole to a cognicise training program on lower-extremity function in community-dwelling older adults with mild cognitive impairment (MCI). In this randomized controlled intervention study, we will recruit 40 community-dwelling individuals aged ≥55 years with MCI. Experimental group (n=20) will receive cognicise training program with insole intervention (6 hours/day), while the control group (n=20) only undergo cognicise training. A 1-h training session will be given three times a week for 12 weeks for both groups. The outcomes include static standing balance, functional reach test, timed-up-and-go test, 10-m obstacle crossing, the Short Physical Performance Battery (SPPB), and gait assessment during single- and dual-task walking for 20 m at self-selected comfortable pace while performing serial subtractions (cognitive interference) or carrying a tray (motor interference). The results of the current study are expected to provide evidences in supporting the use of arch support insole among community-dwelling older adults with MCI. Interventions combing physical-cognitive training and insole for providing mechanical stability and somatosensory stimulation may serve as potential strategies for fall prevention.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 55 years and over; (2) able to walk more than 20 m without walking aids; (3) had a Montreal Cognitive Assessment (MoCA) score lower than 26 ; (4) had self-reported memory complaints; and (5) had the ability to perform ADLs.

Exclusion Criteria:

* (1) dementia; (2) a history of malignant tumors ; (3) the presence of an unstable neurological or orthopedic disease, or visual problems interfering with participation in the study; and (4) an education level less than 6 years (elementary school).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-25 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of static standing balance | at baseline and after 12-wk of intervention
  30-s static standing balance
Change of timed-up-and-go test | at baseline and after 12-wk of intervention
  3-m timed-up-and-go test
Change of 10-m obstacle crossing | at baseline and after 12-wk of intervention
  10-m obstacle crossing
Change of functional reach test | at baseline and after 12-wk of intervention
  functional reach test
Change of Short Physical Performance Battery | at baseline and after 12-wk of intervention
  Short Physical Performance Battery
Change of gait | at baseline and after 12-wk of intervention
  single- and dual-task walking for 20 m at self-selected comfortable pace while performing serial subtractions (cognitive interference) or carrying a tray (motor interference)

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Yi Song, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided